CLINICAL TRIAL: NCT02112019
Title: Endoscopic Treatment of Salivary Glands Affected by Sjögren's Syndrome; A Randomised Controlled Pilot Study
Brief Title: Endoscopic Treatment of Salivary Glands Affected by Sjögren's Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Derk Jan Jager (Other)
Responsible Party: Sponsor-Investigator, Derk Jan Jager, DMD PhD, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NL44018.029.13
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Sjögren's Syndrome
Keywords: Sjögren's Syndrome; Sialoendoscopy; Saliva; Dry Mouth
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia | interventions — Sodium Chloride; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sialoendoscopy with saline (Experimental): By performing a sialoendoscopy, the ducts of the salivary glands are rinsed with saline and possible strictures are dilated
  Interventions: Procedure: Sialoendoscopy; Drug: saline
- Sialoendoscopy: saline and hydrocortisone (Active Comparator): By performing a sialoendoscopy, the ducts of the salivary glands are rinsed with saline and hydrocortisone and possible strictures are dilated
  Interventions: Procedure: Sialoendoscopy; Drug: saline; Drug: hydrocortisone
- Control: no treatment (No Intervention)

INTERVENTIONS:
Procedure: Sialoendoscopy
  Arms: Sialoendoscopy with saline; Sialoendoscopy: saline and hydrocortisone
Drug: saline
  Arms: Sialoendoscopy with saline; Sialoendoscopy: saline and hydrocortisone
Drug: hydrocortisone
  Arms: Sialoendoscopy: saline and hydrocortisone

SUMMARY:
Sjögren's syndrome (SS) is an autoimmune inflammatory disorder of the exocrine glands. It particularly affects the lacrimal and salivary glands. Severe dry mouth and eyes are frequently reported as presenting symptoms. These symptoms are in many cases accompanied by nonspecific symptoms, such as malaise and fatigue. In addition, extraglandular manifestations, like purpura, polyneuropathy, and arthritis, can be present. SS affects mainly women with a female/male ratio of 9:1 and can occur at all ages. Due to the irreversible damage to the saliva producing cells, the quantity and quality of saliva reduces. The progressive nature of the syndrome results in a further reduction of salivary flow. Due to hyposalivation the patients suffer from progressive dental decay, dental erosion, severe dry mouth complaints (i.e. eating and swallowing problems, lack of taste), inflammation of the oral mucosa and lack of retention of removable dentures. Overall, this can be qualified as a reduction in the quality of life. Until now no effective (palliative) therapy to relieve dry mouth complaints is available. A recent case series study suggests that an endoscopic technique (sialoendoscopy) is able to alleviate the symptoms of patients suffering from SS. In this technique the ducts of the salivary glands are rinsed with saline and cortisone and possible strictures are dilated. It is hypothesised that performing a sialoendoscopic treatment will raise or restore (un)stimulated salivary flow levels and improve the reported mouthfeel score.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosed (by the European League Against Rheumatism guidelines) primary or secondary Syndrome of Sjögren
* Age: > 18 years and < 70 years
* A remaining salivary flow

Exclusion Criteria:

* A complete lack of measurable salivary flow, also after stimulation of the glands by taste or chewing
* Acute sialadenitis
* Use of sialogogue medication (i.e. pilocarpine or cevimeline)
* Other severe illnesses or physical conditions that make a treatment under general anesthesia impossible or highly riskful.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change, compared to baseline and to a non-treatment control group, in unstimulated whole mouth saliva in ml/min after sialoendoscopic treatment | Baseline, 2 years
  To determine the change, compared to baseline and to a non-treatment control group, in the unstimulated whole mouth (UWS) salivary flow after performing sialoendoscopic rinsing (with or without hydrocortisone) and dilatation of strictures of the salivary ducts of the major salivary glands.

SECONDARY OUTCOMES:
Change, compared to baseline and to a non-treatment control group, in the stimulated parotid salivary flow after performing sialoendoscopic rinsing (with or without hydrocortisone) | Baseline, 2 years
  Change, compared to baseline and to a non-treatment control group, in the stimulated parotid (SP) salivary flow after performing sialoendoscopic rinsing (with or without hydrocortisone) and dilatation of strictures of the salivary ducts of the major salivary glands.
Change in mouthfeel score (XI score) | Baseline, 2 years
  Change in mouthfeel score (XI score) after sialoendoscopic treatment, with or without rinsing with hydrocortisone, compared to baseline and compared to a non-treatment control group
Change in the EULAR SS Patient Reported Index score | Baseline, 2 years
  Change in the ESSPRI (EULAR SS Patient Reported Index) score after sialoendoscopic treatment, with or without rinsing with hydrocortisone, compared to baseline and compared to a non-treatment control group
Change in the CODS score | Baseline, 2 years
  Change in the CODS score after sialoendoscopic treatment, with or without rinsing with hydrocortisone, compared to baseline and compared to a non-treatment control group

CONTACTS AND LOCATIONS:
Locations (1):
- VU Medical Center department of Maxillofacial surgery, Amsterdam, Netherlands